CLINICAL TRIAL: NCT05837169
Title: Randomized Study with Wait-list Control to Evaluate the Impact of a Stress Reduction Intervention Based on Mindfulness Offered Virtually to Reduce Anxiety Levels in Breast Cancer Survivors
Brief Title: Randomized Study to Evaluate an Intervention Based on Mindfulness to Reduce Anxiety in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicos e Investigadores en la Lucha contra el Cancer de Mama (Other)
Responsible Party: Principal Investigator, Cynthia Villarreal Garza, Principal Investigator, Medicos e Investigadores en la Lucha contra el Cancer de Mama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECA-MIND
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Breast Cancer; Survivorship
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, the study will be open and participants will know which group they belong to. However, the statistician will be blinded in order to reduce the risk of introducing bias when interpreting the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The MBSR program will be offered through the Zoom platform. It consists of a total of 8 weekly sessions, with an approximate duration of 2 hours per session. During these sessions, patients will be instructed in exercises to promote mindfulness, including body awareness (body scan), gentle yoga exercises, and meditation. Additionally, a digital manual will be delivered with exercises that can be done at home, 8 audios with guided exercises and a video with balance and flexibility postures. Patients will be instructed to practice mindfulness exercises at least twice a day, lasting approximately 20 min per exercise, to cultivate the incorporation of meditation into their daily lives.
  Interventions: Other: Mindfulness-based stress reduction
- Wait-list control group (No Intervention)

INTERVENTIONS:
Other: Mindfulness-based stress reduction — The control group will be assessed with the study surveys at baseline, will not receive MBSR intervention for the following 8 weeks, and will subsequently be reassessed with the study surveys at the same time points as the intervention group. At the end of the recruitment and follow-up of all the participants, the study will end and the control group will be able to receive the MBSR intervention free of charge according to the preference of the participants.
  Arms: Intervention group

SUMMARY:
The diagnosis and treatment of breast cancer (BC) can drastically affect the quality of life of patients with this disease by causing symptoms of vasomotor disorders, insomnia, depression and anxiety. Mindfulness-Based Stress Reduction (MBSR) is a program dedicated to fostering complete awareness in the present in order to accept the moment, thereby reducing stress. Previous studies have shown that MBSR benefits patients with chronic conditions such as mood disorders and chronic pain, as well as patients with BC. However, its usefulness in Mexican patients has not been previously studied.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical study, controlled by a wait-list group and blinded to the statistician, with the main objective of evaluating whether an MBSR intervention offered virtually allows reducing the levels of anxiety of BC survivors.

The randomized design will make it possible to compare participants' levels of anxiety, depression, fear of recurrence, and physical symptoms according to whether they participate in a virtual MBSR program or do not. In addition, the randomized design will reduce the possible impact of confounding variables, facilitating direct comparison between the two groups.

Invitation to the study will be made through social networks of Mexican civil associations and through the dissemination of the study by specialists in oncology. It will be done this way because the intervention through an online mindfulness program can be delivered to a considerable volume of BC survivors with internet access, regardless of their place of residence or medical care.

Participants will be assigned to the intervention group or the wait-list control group. Those randomized to the control group will not receive the MBSR intervention during the study period, while those randomized to the intervention group will participate in a virtual MBSR program, which is described below. A wait-list control group will be used with the aim that all participants have the opportunity to receive the MBSR intervention and at the same time allow comparison of the effect of the program with a group without intervention. Given that anxiety has a significant negative impact on people's well-being, it is appropriate to offer the control group the possibility of receiving an intervention if its effectiveness is demonstrated. The control group will be assessed with the study surveys at baseline, will not receive MBSR intervention for the following 8 weeks, and will subsequently be reassessed with the study surveys at the same time points as the intervention group. At the end of the recruitment and follow-up of all the participants, the study will end and the control group will be able to receive the MBSR intervention free of charge according to the preference of the participants.

BC survivors will be invited to participate through an electronic link with a selection questionnaire asking about the inclusion and exclusion criteria. In particular, the General Anxiety Disorder-7 (GAD-7) tool will allow for anxiety screening in order to determine if those interested in participating have the minimum level of anxiety required to be included in the study. Through that same electronic link, those who meet the eligibility criteria will be invited to read and sign the electronic informed consent. Those who accept will be randomly assigned to the intervention group or control group, in a 1:1 ratio considering a stratification according to the severity of anxiety measured by GAD-7 (moderate vs. severe) and menopausal status (pre- vs. post-menopause) in the questionnaire. of selection. Likewise, they will be asked for contact information (i.e., telephone and email) in order to send them the study surveys (participants in both groups) and the electronic links for the MBSR program sessions (participants in the intervention group). At this baseline time (T1), participants randomized to either group will answer the study surveys to assess symptoms of anxiety, depression, and fatigue.

Subsequently, the intervention group will participate in the online MBSR intervention for 8 weeks, while the control group will be registered on a waiting list and will be able to receive the intervention once the study is finished. For both the intervention group and the control group, the online MBSR program will be offered free of charge.

Participants will answer the study surveys again 1 week (T2), 3 months (T3) and 6 months (T4) after completing the online mindfulness program. In the case of participants randomized to the control group, these times correspond to 9 weeks (T2), 5 months (T3) and 8 months (T4) of follow-up. Additionally, in T2 the participants randomized to the intervention group will answer a satisfaction survey with the online MBSR program. At the end of the recruitment and follow-up of the participants, the study will end and those randomized to the control group by waiting list will be able to receive the MBSR intervention online if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 0-III BC
* Between 1 and 5 years after receiving the diagnosis of BC
* Not being treated with chemotherapy or radiotherapy during the duration of the study
* Score ≥10 on the GAD-7 tool (moderate to severe anxiety)
* Internet access at home
* Availability to participate in the MBSR intervention virtually for 8 weeks
* Availability to answer the follow-up questionnaires during the duration of the study

Exclusion Criteria:

* Metastatic disease
* Score <10 on the GAD-7 tool (mild anxiety)
* Current meditation practice
* Inability to read or write

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Anxiety | 8 months
  Anxiety level, as measured by the General Anxiety Disorder-7 (GAD-7) tool. GAD-7 is a validated tool made up of 7 items that are each rated from 0-3, thus the total score can range from 0-21. A score between 10-14 suggests moderate anxiety and a score of 15-21 suggests severe anxiety. Therefore, a score ≥10 has been established as cut-off point to identify cases of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrigno Guajardo A, Salazar-Alejo M, Mesa-Chavez F, Gutierrez-Ornelas J, Platas A, Verduzco-Aguirre H, Villarreal-Garza C. Effectiveness of an online mindfulness-based stress-reduction intervention to reduce anxiety in breast cancer survivors: a randomized-controlled trial. Support Care Cancer. 2025 Jun 24;33(7):623. doi: 10.1007/s00520-025-09681-6. PMID 40555874